CLINICAL TRIAL: NCT04768920
Title: Examining Feasibility and Acceptability of Telemedicine for Substance Use Disorder (SUD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Allison Lin, Assistant Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00189259
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Substance Use Disorders; Substance Use; Substance Dependence
Keywords: Telehealth; Motivational interviewing; Cognitive behavioral therapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teletx (Experimental): The evidence-based manualized psychosocial programs that will be delivered via telehealth are adaptations of cognitive behavioral therapy, motivational interviewing, and other psychosocial interventions to enhance initial and ongoing treatment engagement. TeleTx consists of up to 8 ~30-50 minute psychosocial sessions delivered via phone or videoconference platform (e.g. Zoom etc).
  Interventions: Behavioral: MI-CBT Teletx

INTERVENTIONS:
Behavioral: MI-CBT Teletx — Participants will first receive a 20-45 min phone or video session focused on raising participants' motivation to engage in treatment activities and psychoeducation material about substance use (i.e. "engagement session") including possible discussion about risks of substance use, value of alternative healthier activities, and the community and crisis resources pamphlet. The evidence-based manualized psychosocial programs that will be delivered via telehealth are adaptations of cognitive behavioral therapy, motivational interviewing, and other psychosocial interventions to enhance initial and ongoing treatment engagement. TeleTx consists of up to 8 ~30-50 minute psychosocial sessions delivered via phone or videoconference platform (e.g. Zoom etc)

SUMMARY:
The objective of this pilot intervention study is to iteratively refine motivational interviewing and psychosocial intervention programs delivered via telehealth (Teletx) to help improve substance use and other related outcomes in SUD patients who are not receiving SUD care. We will examine feasibility and acceptability of these pilot psychosocial programs in a total of n=50 participants. The goal is to refine the programs to improve acceptability and feasibility and collect preliminary data for a future fully powered randomized controlled trial (RCT) in the future.

In addition to study sessions, participants that are enrolled in the study will complete surveys prior to, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient care at Michigan Medicine in past year
* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) SUD diagnosis and/or substance use on average of 2 days a week over the past month
* Have a Smart phone, tablet or another Wi-Fi or data-enabled device (e.g. with a camera)

Exclusion Criteria:

* Inability to speak or understand English
* Conditions that preclude informed consent (e.g., acute psychosis, cognitive deficits) or understanding of assessment or program content
* Prior alcohol withdrawal seizures or delirium tremens (DTs). Those who are at-risk of complicated withdrawal (e.g., seizures, DTs) require greater medical attention and will be excluded and referred to their clinician for medical management.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention (engagement) | 8 weeks
  Percent (%) of participants engaging in the intervention
Tele-Tx Intervention acceptability | 8 weeks
  Study-specific acceptability rating completed by participants. Based on Likert scale, higher scores indicate greater treatment acceptability

OTHER OUTCOMES:
Change in frequency of substance use as reported on the Timeline Follow-Back (TLFB) | baseline, 8 weeks post-baseline
  Based on frequency and quantity, higher scores indicate worse outcome.
Change in Alcohol Consumption | baseline, 8 weeks post baseline
  Alcohol consumption will be assessed using the 30-day Timeline Follow-Back (TLFB). The TLFB will capture information on the frequency and quantity of alcohol use including binge drinking, with total consumption calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No